CLINICAL TRIAL: NCT04088526
Title: Survey and Reduction of Mortality in Uremic Patients During Peridialysis Period Via Intervention of Risk Factors
Brief Title: Survey and Reduction of Mortality in Peridialysis Uremic Patients Via Intervention of Risk Factors
Acronym: SURVIVOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Changlin Mei, Director of Kidney Institution of PLA, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CZKIPLA-ESRD-001
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Through the effective intervention of risk factors for death in patients with dialysis, the effect of mortality of peri-dialysis patients was observed.
  Interventions: Combination Product: intervention group

INTERVENTIONS:
Combination Product: intervention group — Through effective intervention combined with drugs and dietary guidance within 3 to 6 months, all the observation markers including blood pressure and laboratory results will reach the target target value.

SUMMARY:
In patients with non-dialysis-dependent end stage kidney disease (ESKD) the common transition of care to renal replacement therapy is dialysis. Each year over 70 000 Chinese transition from non-dialysis-dependent ESKD to dialysis. Whereas dialysis therapy is intended to be life-sustaining, ESKD patients have a 10-fold or higher risk of death compared with the general population. Mortality rates are even higher upon transition and in the first year, especially in the first 3 to 6 months following the transition to dialysis, yet it remains unknown which is the contributing cause of this high death rate. Hence, there is an urgent need to examine the emerging field of Transition of Care in ESKD. We suggest the term "peridialysis period" for this transition period for ESKD patients, so that the transition of care from non-dialysis-dependent ESKD to dialysis ESKD can be more pragmatically defined and studied. In the current study, we will investigate the mortality and its risk factors of ESKD patients during peridialysis period, and improve the survival rate and quality of life of peridialysis ESKD patients by intervening the risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with end stage kidney disease (eGFR<15ml/min/1.73m2) or newly started dialysis with 3 months at all hospitals in Yangzhou, China since January 1, 2016

Exclusion Criteria:

* Patients who have had a history of dialysis and have been transferred to Yangzhou during this period;
* patients who are transferred to a dialysis area outside Yangzhou City
* Patients who give up dialysis treatment
* patient whose renal function recover and stop dialysis treatment;
* Patient who receive kidney transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | one year
  mortality and death cause

SECONDARY OUTCOMES:
hospitalization | one year
  hospitalization rate and cause

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, M.D., Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Department of Nephrology, Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China